CLINICAL TRIAL: NCT01784198
Title: Determination of Protein Requirements in Healthy Pregnant Women Using Indicator Amino Acid Oxidation Technique
Brief Title: Determination of Protein Requirements in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H11-00070
Record Dates: First submitted 2013-01-17; First posted 2013-02-05 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pregnancy
Keywords: pregnancy; protein requirements; Indicator Amino acid oxidation; Stable isotopes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Protein Intake (Experimental): Dietary supplement:Protein intake
  Interventions: Dietary Supplement: Protein Intake

INTERVENTIONS:
Dietary Supplement: Protein Intake — Oral consumption of Eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.

SUMMARY:
Protein is an essential part of our diet. It is used to build muscle and body tissue, send signals throughout our body and to support the immune system. Dietary protein is even more crucial during pregnancy as it is needed for healthy growth and development of the baby. There is very minimal data available on how much additional protein is required during pregnancy. Current recommendations are based on older techniques such as nitrogen balance studies of non-pregnant adults and minimally based on pregnancy specific data. There is no scientific information regarding the amount of protein needed during different stages of pregnancy.

The investigators hypothesize that the current recommendations of protein intake during pregnancy are underestimated.

The goal of this study is to measure protein requirement in healthy pregnant women (19-35y)using a more quick and modern technique called the indicator amino acid oxidation technique (IAAO).

ELIGIBILITY:
Inclusion Criteria:Healthy pregnant women

* Singleton pregnancy
* Maternal age 19-35y
* In good health (free of chronic/acute disease,full range of physical mobility)
* Healthy pre-pregnancy body mass index

Exclusion Criteria:Women

* not pregnant
* Pregnant with more than one child
* Singleton pregnancy outside the age range of 19-35y
* Not in good health or have a metabolic, neurological, genetic, or immune disorder, including gestational diabetes or anemia
* smoke or consume alcohol during their pregnancy
* classified as underweight (<18.5 kg/m2), overweight (25-30 kg/m2) or obese (>30 kg/m2)
* allergic to eggs and egg protein
* severe nausea/vomiting throughout their pregnancy

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
13 Carbon dioxide production | 8 hours (1 study day)
  Urine and breath samples will be collected during the study to measure the rate of oxidation of tracer in expired breath and flux by enrichment in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — Child & Family Research Institute/University of British Columbia
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Stephens TV, Payne M, Ball RO, Pencharz PB, Elango R. Protein requirements of healthy pregnant women during early and late gestation are higher than current recommendations. J Nutr. 2015 Jan;145(1):73-8. doi: 10.3945/jn.114.198622. Epub 2014 Sep 24. PMID 25527661